CLINICAL TRIAL: NCT01697501
Title: Cross-sectional Multicenter Study Evaluating the IL28B Polymorphism in Patients With HBeAg-negative Chronic Hepatitis B Treated With Pegylated Interferon Alfa-2a in the Course of Peg.Be.Liver Study
Brief Title: A Study Evaluating IL28B Polymorphism in Patients With HBeAg-Negative Chronic Hepatitis B Treated With Pegasys (Peginterferon Alfa-2a) in Study ML18253
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ML28470; 2012-002777-56 (EudraCT Number)
Record Dates: First submitted 2012-09-28; First posted 2012-10-02 (Estimated); Results first posted 2015-07-10 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2017-03

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic

ARMS (1):
- Chronic hepatitis B patients (Experimental)
  Interventions: Other: Interleukin 28B testing

INTERVENTIONS:
Other: Interleukin 28B testing — Blood sampling for IL28B genotyping

SUMMARY:
This cross-sectional multicenter study will evaluate the IL28B polymorphism in patients with HBeAg-negative chronic hepatitis B treated with Pegasys (peginterferon alfa-2a) in the predecessor ML18253 study. The study consists of a single visit where eligible patients will undergo a blood test for IL28B genotyping, with a phone follow-up 7 days after the visit.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Chronic hepatitis B
* Previous participation in study ML18253
* Administration of at least one dose of the study drug during ML18253 study

Exclusion Criteria:

* Patients not satisfying the above inclusion criteria will not be enrolled in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2012-11-08 (Actual); Primary Completion 2013-06-21 (Actual); Study Completion 2013-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (12):
- Italy (12):
  - Azienda Ospedaliera Policlinico Consorziale di Bari; Clinica Malattie Infettive, Bari, Apulia
  - Ospedale de Bellis; Reparto Medicina Generale, Castellana Grotte, Apulia
  - Az. Osp. S. Sebastiano; Divisione Malattie Infettive, Caserta, Campania
  - Az. Osp. Cardarelli; Unita Operativa A Struttura Complessa Di Epatologia, Napoli, Campania
  - UNI DEGLI STUDI - POLICLINICA S. ORSOLA; Dipartimento Malattie dell'Apparato Digerente e Medicina In, Bologna, Emilia-Romagna
  - Az. Osp. Uni Ria Di Parma; Gastro-Enterology, Parma, Emilia-Romagna
  - Fondazione IRCCS Ospedale Maggiore Policlinico; Gastroenterologia, Milan, Lombardy
  - Ospedale Maggiore Policlinico; Iii Divisione Medicina Generale, Milan, Lombardy
  - Uni Di Cagliari; Dept. Di Scienze Mediche, Cagliari, Sardinia
  - Istituto Di Clinica Medica 1 A; Divisione Di Medicina Generale E Gastroenterologia, Palermo, Sicily
  - Ospedale Cisanello - Az. Osp. Pisana; Unità Operativa Di Gastroenterologia Ed Epatologia, Pisa, Tuscany
  - Az. Osp. Di Padova; Dipart. Scienze Chirurgiche E Gastroent., Padua, Veneto

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants in the safety analysis set included 88 patients with HBeAg-negative chronic hepatitis B enrolled at 12 study centers in Italy.
Pre-assignment Details: Participants in the full analysis set included 86 previously enrolled in the predecessor study ML18253 (NCT01095835), during which they were treated.
Period: Overall Study
Arm/Group | Chronic Hepatitis B Patients
Started | 88
Completed | 86
Not Completed | 2
Not completed — Protocol Violation | 2

BASELINE CHARACTERISTICS:
Arm/Group | Chronic Hepatitis B Patients
Number analyzed (Participants) | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.7 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 65

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Viral Response (SVR) Defined as HBV DNA ≤ 2000 IU/ml at IL28B Genotype rs12979860 at End of Follow-up (EoF)
Time Frame: EoF, as defined in the predecessor study, was at 48 weeks after the end of treatment.
Population: Full analysis set (FAS), defined as all subjects who completed
Measure: Number; unit: percentage of participants
Groups:
- "CC"; "TC"; "TT"; "TC+TT"; "Overall": at IL28B genotype rs12979860
Arm/Group | "CC" | "TC" | "TT" | "TC+TT" | "Overall"
Number analyzed (Participants) | 35 | 41 | 10 | 51 | 86
percentage of participants | 20.0 | 17.1 | 20.0 | 17.6 | 18.6
Statistical Analysis 1: Comparison: "CC" vs "TC+TT"; Test type: Superiority or Other; p = 0.7831, univariate logistic analysis; Odds Ratio (OR) = 0.86, 95% CI 2-sided [0.29 to 2.57]

2. Primary Outcome: Percentage of Participants With SVR Defined as HBV DNA ≤ 2000 IU/ml at IL28B Genotype rs8099917 at EoF
Time Frame: EoF
Population: FAS
Measure: Number; unit: percentage of participants
Groups:
- "TT"; "GT"; "GG"; "GT+GG"; "Overall": at IL28B genotype rs8099917
Arm/Group | "TT" | "GT" | "GG" | "GT+GG" | "Overall"
Number analyzed (Participants) | 52 | 31 | 3 | 34 | 86
percentage of participants | 23.1 | 12.9 | 0.0 | 11.8 | 18.6
Statistical Analysis 1: Comparison: "TT" vs "GT+GG"; Test type: Superiority or Other; p = 0.1951, univariate logistic analysis; Odds Ratio (OR) = 2.25, 95% CI 2-sided [0.66 to 7.67]

3. Secondary Outcome: Percentage of Participants With HBV DNA ≤ 2000 IU/ml at IL28B Genotype rs12979860 at End of Treatment (EoT)
Time Frame: EoT, as defined in the predecessor study, was at Week 48 or Week 96
Population: Full analysis set (FAS), defined as all subjects who completed
Measure: Number; unit: percentage of participants
Arm/Group | "CC" | "TC" | "TT" | "TC+TT" | "Overall"
Number analyzed (Participants) | 35 | 41 | 10 | 51 | 86
percentage of participants | 74.3 | 65.9 | 50.0 | 62.7 | 67.4
Statistical Analysis 1: Comparison: "TC" vs "TC+TT"; Test type: Superiority or Other; p = 0.2642, Wald Chi Square

4. Secondary Outcome: Percentage of Participants With HBV DNA ≤ 2000 IU/ml at IL28B Genotype rs8099917 at EoT
Time Frame: EoT
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | "TT" | "GT" | "GG" | "GT+GG" | "Overall"
Number analyzed (Participants) | 52 | 31 | 3 | 34 | 86
percentage of participants | 75.0 | 54.8 | 66.7 | 55.9 | 67.4
Statistical Analysis 1: Comparison: "TT" vs "GT+GG"; Test type: Superiority or Other; p = 0.0672, Wald Chi Square

5. Secondary Outcome: Percentage of Participants With HBsAg < 0.05 IU/ml at IL28B Genotype rs12979860 at EoT and EoF
Time Frame: EoT and EoF
Population: Full analysis set (FAS), defined as all subjects who completed
Measure: Number; unit: percentage of participants
Arm/Group | "CC" | "TC" | "TT" | "TC+TT" | "Overall"
Number analyzed (Participants) | 35 | 41 | 10 | 51 | 86
percentage of participants
  EoT | 2.9 | 2.4 | 0.0 | 2.0 | 2.3
  EoF | 0.0 | 4.9 | 0.0 | 3.9 | 2.3

6. Secondary Outcome: Percentage of Participants With HBsAg < 0.05 IU/ml at IL28B Genotype rs8099917 at EoT and EoF
Time Frame: EoT and EoF
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | "TT" | "GT" | "GG" | "GT+GG" | "Overall"
Number analyzed (Participants) | 52 | 31 | 3 | 34 | 86
percentage of participants
  EoT | 3.8 | 0.0 | 0.0 | 0.0 | 2.3
  EoF | 3.8 | 0.0 | 0.0 | 0.0 | 2.3

7. Secondary Outcome: Percentage of Participants With HBsAg ≤ 10 IU/ml at IL28B Genotype rs12979860 at EoT and EoF
Time Frame: EoT and EoF
Population: Full analysis set (FAS), defined as all subjects who completed
Measure: Number; unit: percentage of participants
Arm/Group | "CC" | "TC" | "TT" | "TC+TT" | "Overall"
Number analyzed (Participants) | 35 | 41 | 10 | 51 | 86
percentage of participants
  EoT | 8.6 | 7.3 | 0.0 | 5.9 | 7.0
  EoF | 2.9 | 4.9 | 0.0 | 3.9 | 3.5

8. Secondary Outcome: Percentage of Participants With HBsAg ≤ 10 IU/ml at IL28B Genotype rs8099917 at EoT and EoF
Time Frame: EoT and EoF
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | "TT" | "GT" | "GG" | "GT+GG" | "Overall"
Number analyzed (Participants) | 52 | 31 | 3 | 34 | 86
percentage of participants
  EoT | 11.5 | 0.0 | 0.0 | 0.0 | 7.0
  EoF | 5.8 | 0.0 | 0.0 | 0.0 | 3.5

ADVERSE EVENTS:
Time Frame: The study consisted of a single visit where eligible patients undergo a blood test for IL28B genotyping, with a phone follow-up 7 days after the visit. All subjects enrolled are included in the safety analysis set.
Description: Adverse events were to be reported on a per subject basis by severity and relationship to study procedures.
Arm/Group | Chronic Hepatitis B Patients
Serious Adverse Events (participants affected / at risk) | 0/88
Other Adverse Events (participants affected / at risk) | 0/88

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.